CLINICAL TRIAL: NCT05885698
Title: Molecularly Informed Lung Cancer Treatment in a Community Cancer Network: A Longitudinal Prospective RWE Study (MYLUNG Consortium Part 3: Observational Study)
Brief Title: MYLUNG Consortium Part 3: Observational Study
Acronym: MYLUNG
Status: Recruiting | Type: Observational
Sponsor: US Oncology Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 22285
Record Dates: First submitted 2023-02-22; First posted 2023-06-02 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Lung Cancer; Squamous Non-small Cell Lung Cancer; Non-squamous Non-small Cell Lung Cancer; Biomarker Testing; Tumor Tissue Testing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-small Cell Lung Cancer

SUMMARY:
This longitudinal study looks to quantify the testing timeline, operational barriers, and outcomes of biomarker-guided therapy in a large, community-based, and largely unselected patient population with early stage and advanced stage, treatment-naive non-small cell lung cancer, whether squamous or non-squamous.

DETAILED DESCRIPTION:
Lung cancer remains the most lethal malignancy in men and women in the U.S. Providing high quality management of these patients in the community setting as compared to hospital or academic centers offers the opportunity to reduce cost without sacrificing clinical outcome and simultaneously improving patient convenience and value. Many patients diagnosed with late-stage cancers can benefit from advanced biomarker testing, yet not all eligible patients receive this type of diagnostic testing today.

Within advanced non-small-cell lung cancer (aNSCLC), there are many specific somatic mutations observed in select patient populations that have targeted highly effective and less toxic therapies. National guidelines have advocated for broad tumor molecular profiling as a part of the standard diagnostic evaluation for aNSCLC, with the goal of identifying driver mutations for which effective therapies or clinical trials are available.

Furthermore, there is emerging evidence that molecular testing can impact treatment choices in earlier stages of lung cancer. However, adherence to genomic testing guidelines presents unique challenges to community oncologists. While most oncology clinical research has been conducted at well-established academic medical centers, over 85% of cancer patients are diagnosed and treated at local, community-based clinical practices. Barriers exist in the ability to order these tests efficiently, in a timely manner, and reimbursed accordingly. Furthermore, patient care can vary drastically based on community-associated disparities.

This longitudinal clinical trial will generate Real World Evidence (RWE) to validate efficacy of first treatment regimen in newly diagnosed patients with non-small cell lung cancer. The MYLUNG Program integrates three separate protocols: Protocol #1 interrogated historical data from a large number of practices seeing lung cancer patients to evaluate biomarker testing, decision making patterns, the patient journey, and the tissue journey; Protocol #2 prospectively evaluated the patient journey in a limited number of index practices focused on testing; integration of testing results; and treatments. Interventional strategies to optimize these objectives will be developed and integrated into various interventions all aimed at improving biomarker testing rates. Protocol #3 (22285) will serve as a resource to monitor the impact of these strategies on the patient journey as it relates to shared decision making, and will continue to prospectively evaluate the patient journey in a limited number of index practices focused on testing, integration of testing results and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years and older) with newly diagnosed early stage, locally advanced or metastatic non-small cell lung cancer
* Must be eligible for systemic therapy based on the treating provider's assessment. If systemic therapy was recommended and documented by the treating provider but the patient declined, they can still be eligible for the study. Patients can be enrolled prior to start of treatment.
* Subjects who developed locally advanced or metastatic disease after receiving adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of locally advanced or metastatic disease
* Subjects must be enrolled within 30 days of initiation of systemic therapy
* Signed informed consent

Exclusion Criteria:

* Stage IA at the time of enrollment
* Subjects with small cell lung cancer
* Subjects with Unknown primary tumor origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This longitudinal study looks to quantify the testing timeline, operational barriers, and outcomes of biomarker-guided therapy in a large, community-based, and largely unselected patient population with early stage and advanced stage, treatment naive non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Who Receive Biomarker Test Results Prior to Systemic Therapy or Death | 5 years from date of enrollment into study
Proportion of Patients Who Receive Single-gene Testing Compared to Those that Receive Comprehensive Biomarker Testing | 5 years from date of enrollment into study
  Comprehensive biomarker testing is defined as both PD-L1 testing to guide the use of immunotherapies and testing for all genomic alterations for which there are FDA-approved therapies including (but not limited to) EGFR, ALK, ROS1, BRAF, NTRK, RET, KRAS and MET.
For Patients without Biomarker Test Results, List Reasons for Not Conducting Testing | 5 years from date of enrollment into study
  1. Clinical deterioration, clinical crisis
  2. Tissue: obtaining sample, tissue retrieval
  3. Assay failure for 1 or more biomarkers: Quantity Not Sufficient (QNS), Quality Assurance (QA) fail, test failure
  4. Patient/provider attitudes & perceptions
  5. Provider knowledge about testing options
  6. Patient knowledge about biomarker testing
  7. Payor Coverage: prior authorization denial, payor refusal
  8. Financial barriers: uncovered costs, reimbursement

SECONDARY OUTCOMES:
Proportion of patients placed on biomarker-directed first treatment regimen vs those who were not | 5 years from date of enrollment into study
Time span between first systemic therapy as compared to date of initial presentation, date of diagnostic biopsy, date of first visit to a medical oncologist, and date of biomarker test order(s) and result(s). | 5 years from date of enrollment into study
For Patients who Receive Comprehensive Biomarker Testing, list Types of Test Ordered | 5 years from date of enrollment into study
For Patients without Biomarker-Directed First Treatment Regimen, Catalog Reasons for Not Prescribing Biomarker-Targeted Therapy | 5 years from date of enrollment into study
  For patients who have received biomarker test results with at least one actionable mutation, catalog the reason for not prescribing biomarker-targeted therapy.
  1. Lack of availability or delays in obtaining targeted therapy
  2. Misinterpretation of test results
  3. Clinical contraindications (allergies, end organ dysfunction, active autoimmune disease, etc.)
  4. Patient/provider attitudes and perceptions
  5. Financial barriers / Uncovered costs
  6. Patient performance status
For Patients who Receive Comprehensive Biomarker Testing, list Types of Resulting Treatment Regimen Assigned | 5 years from date of enrollment into study
Characteristics of Cancer Care Practices: Number of Geographic Clinical Locations Per Practice | 5 years from date of enrollment into study
Characteristics of Cancer Care Practices: Rural Setting vs Urban Setting at each Practice | 5 years from date of enrollment into study
Characteristics of Cancer Care Practices: Number of Staff per Practice | 5 years from date of enrollment into study
Characteristics of Cancer Care Practices: Patient Volume per Practice | 5 years from date of enrollment into study

CONTACTS AND LOCATIONS:
Overall Officials: Makenzi C. Evangelist, MD, Principal Investigator — New York Oncology Hematology; Patrick J. Ward, MD, Principal Investigator — Oncology Hematology Care Clinical Trials, LLC
Locations (17):
- United States (17):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Arizona Oncology Associates, PC - NAHOA, Prescott Valley, Arizona
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - New York Oncology Hematology, P.C., Albany, New York
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington